CLINICAL TRIAL: NCT07376252
Title: Development and Evaluation of a Mobile Health Application (APP) Aimed at Parents for the Prevention of Overweight and Obesity in School Children in Mexico City. Apply for Your Health!
Brief Title: Use of a Mobile Application by Parents to Prevent Obesity in Their Children Apply for Your Health
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Infantil de Mexico Federico Gomez (Other)
Collaborators: Secretaría de Educación, Ciencia, Tecnología e Innovación de la Ciudad de México (Unknown); Fundación Gonzalo Río Arronte (Unknown)
Responsible Party: Principal Investigator, Jenny Vilchis Gil, Dr., Hospital Infantil de Mexico Federico Gomez
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: HIM 2017-086
Record Dates: First submitted 2026-01-22; First posted 2026-01-29 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Obesity; Overweight
Keywords: Obesity; Overweight; schoolchildren; mobile application; eHealth
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Intervention Model Description: In this crossover study, the four schools were randomly assigned to receive the intervention or to be part of the control group. In the second period, the group initially assigned as the control received the intervention, while the group that had received the intervention in the first period did not receive it during this second phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention with the mobile application (Experimental): The educational intervention was implemented through the mobile application "Applícate por tu salud" (Get Healthy), with the goal of sending information to parents on how to improve eating habits at breakfast and school lunch. To this end, recipes, text messages, and infographics related to these topics were developed.
  Interventions: Behavioral: Applícate por tu salud
- Control group (No Intervention): The control group received no educational intervention. Only anthropometric measurements and data collection on diet and physical activity were carried out. However, the results of the anthropometric measurements were given to the parents at different times.

INTERVENTIONS:
Behavioral: Applícate por tu salud — The educational intervention using the mobile application "Applícate por tu salud" aims to promote, improve, and reinforce families' eating habits, focusing on breakfast and school lunches, in order to prevent overweight and obesity in schoolchildren.
  Through the application, using push notifications, tips in the form of text messages, infographics, videos, and recipes are sent four times a week, encouraging positive changes in eating habits related to breakfast and school snacks. The information was formatted as follows: no more than 30 words, suggesting activities that families could implement at home. Eighty-four messages were generated for breakfast and 104 messages for school snacks, including detailed information on planning, selecting, and comparing foods, as well as their preparation and consumption.
  The information was generated by three nutrition experts to standardize the language, and a designer created the infographics, videos, and recipes.
  Arms: Intervention with the mobile application

SUMMARY:
Background. Lifestyles that promote a positive energy balance increase the prevalence of obesity. Due to the magnitude of this problem, community-level strategies are required on how to provide families with useful information to prevent it. Electronic media such as the Internet and mobile health applications are tools that have opened a new audience to send information, they are accessible and powerful, as well as the capacity to reduce associated costs, their access to information is uninterrupted, support , and personalized feedback. There is a need to develop and evaluate mobile health applications to establish consistent and effective methods to produce changes in health behavior in the population.

Aim. To evaluate the impact of a mobile health application in nutrition and physical activity on nutritional status in school children.

Methods. Community essay. Children from 4 primary schools in Mexico City will participate in the educational intervention. The schools were randomly assigned to one of two groups: 1) Apply for your health! group and 2) Control group. The educational intervention through the application will last 12 months and will focus on promoting healthy eating habits and physical activity, empowering parents to change habits. In the second year, the control group will be given access to the mobile application. At baseline, 6, 12, 18 and 24 months, children in both groups will have their nutritional status (anthropometry) and breakfast and school snack habits measured. Statistic analysis. Mixed effects models will be used to evaluate changes in BMI z-score within and between groups.

ELIGIBILITY:
Inclusion Criteria:

1. School-aged children of both sexes, 5-11 years old, enrolled in the selected primary schools.
2. Children and parents who sign the written informed consent and assent form.

Exclusion Criteria:

1. Children participating in any weight loss program, with or without pharmacological treatment.
2. Children with a rheumatological disease, diabetes, thyroid disorder, or any condition that compromises their nutritional status.

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 743 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2024-06-14 (Actual); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
BMI Z-score | Anthropometric evaluations to obtain the BMI Z score are performed at baseline, 6, 12, 18 and 24 months.
  The BMI Z-score variable will be assessed continuously. To evaluate the change in the BMI Z-score, the difference between the corresponding measurements at 6, 12, 18, and 24 months versus the baseline measurement will be calculated.
  A minimum and maximum of -5 to +5 SD will be considered. Likewise, a value closer to zero will be considered the best nutritional condition.

SECONDARY OUTCOMES:
Improvement in the quality of food consumed at breakfast | Information on school breakfasts is collected at baseline, 6, 12, 18 and 24 months
  The change in the quality of food and beverages consumed by students for breakfast before going to school will be evaluated. Information will be collected in two ways: first, students will be asked directly what they ate for breakfast on the day the anthropometric measurements are taken. The foods and beverages consumed will be recorded in portion sizes, as well as whether or not they are ultra-processed.
  Second, a record will be sent to parents via the student so they can note what the student ate for breakfast on the day the anthropometric measurements were taken.
Improvement in the quality of food consumed at school lunch | Information on school lunch is collected at baseline, 6, 12, 18 and 24 months within schools
  The study will evaluate changes in the quality of food and beverages students bring in their school lunches-that is, the food and drinks children bring from home to consume at school. To gather this information, on the day anthropometric measurements are taken at school, children are asked to allow us to record the food and beverages they bring in their lunchboxes. Previously trained and standardized nutritionists will record the food and beverages, including portion sizes, brands, and ultra-processed foods.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Infantil de México Federico Gómez, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: El enlace proporcionado dirige directamente a la página de descarga de la aplicación en la tienda oficial de iOS (App Store), facilitando así el acceso inmediato para los usuarios de dispositivos Apple que deseen instalarla. — https://apps.apple.com/mx/app/appl%C3%ADcate-por-tu-salud/id6451136409
- See also: El enlace proporcionado dirige directamente a la página de descarga de la aplicación en la tienda oficial de ANDORID, facilitando así el acceso inmediato para los usuarios de dispositivos Apple que deseen instalarla. — https://play.google.com/store/apps/details?id=branded.mca07159fbb2c4877a273587ee316dbb9.viviendosaludable&pli=1